CLINICAL TRIAL: NCT05699187
Title: Face Transplantation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrollment
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Curtis L. Cetrulo, MD, Curtis L. Cetrulo, Jr., M.D., FACS, FAAP, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021P002531
Record Dates: First submitted 2023-01-12; First posted 2023-01-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Facial Trauma; Facial Deformity; Facial Injuries
Keywords: Transplant; Face Transplant
MeSH Terms: conditions — Facial Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Face Transplant Recipient (Experimental): The procedure will be carried out simultaneously by two teams of transplant surgeons for each face transplanted in the operation. The teams will be divided between the functions of tissue recovery (donor operation) and transplant surgery (recipient operation). In most cases the facial graft will include the entire nose; the soft tissues of the mid-face, including all its blood vessels, muscles, and nerves; and a significant portion of the mid-facial skeleton.
  Interventions: Procedure: Face allotransplantation

INTERVENTIONS:
Procedure: Face allotransplantation — Facial allotransplantation

SUMMARY:
Face allotransplantation will be performed in facial trauma patients. Immune suppression will primarily be provided according to standard three-drug regimen. The primary outcome to be evaluated in the proposed trial is face allograft acceptance.

DETAILED DESCRIPTION:
Patients with severe facial disfigurement referred or self-identified to the MGH Face Transplantation Program will undergo a consultation with the PI (Dr. Cetrulo) who will perform a thorough clinical assessment and explain in detail the treatment protocol, risks and benefits of the face allotransplantation procedure and alternative options. At the time of appointment, candidates will be first requested to sign a face transplant Research Informed Consent form . Following the signing of these documents, the candidate will meet with the MGH Transplant Center team (see below for description of entire team), a clinical pharmacist, dietician, and a transplant social worker.

Appropriate subjects will then undergo further evaluation/medical screening procedures to determine their candidacy for face transplantation. Prospective recipients who are selected based on results of screening procedures will be invited to review and sign the full informed consent form prior to being wait-listed for the procedure.

There is a significant evaluation using tests, procedures, consults, and evaluations that will be performed as part of the standard of care for those clinically-approved for organ transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Recent (≥6 months) or remote (i.e., several decades) severe facial disfigurement and/or facial functional impairment covering at least 25% of face and/or a major part e.g. nose, lips and desiring face transplantation.
* Aged 18-65 years. Noted should be that the maximal age difference between donor and recipient will be 10 years.
* Completion of the protocol informed consent form.
* No co-existing medical condition which, in the opinion of the study team, could affect the immunomodulatory protocol, surgical procedure, or functional results (see Donor and Recipient Exclusion Criteria below. If the condition is amenable to treatment, the study team must agree that said condition should not significantly enhance the surgical risks of facial transplantation.)
* No co-existing psycho-social problems (i.e., alcoholism, drug abuse).
* Negative for malignancy for past 5 years.
* Negative for HIV at transplant.
* Negative crossmatch with donor.
* If female of child-bearing potential, negative serum pregnancy test. If female of child-bearing potential, consent to use reliable contraception for at least one year following transplantation.
* Patient agrees to comply with the protocol and states a dedication to the immunomodulatory treatment regimen.
* No smoking for 6 months prior to transplant, as confirmed by blood testing.

Exclusion Criteria:

* Positive for any of the following conditions: Untreated sepsis, HIV (active or seropositive), active tuberculosis, hepatitis B or C (HCV Ab+ and HCV RNA+ (HCV Ab+ but RNA negative is acceptable), HBVcAb+, HBVsAg+ or viral DNA+), viral encephalitis, toxoplasmosis, malignancy (within past 5 years), current/recent (within months of donation/consent) IV drug abuse, paralysis of ischemic or traumatic origin, inherited peripheral neuropathy, infectious, post infectious, or inflammatory (axonal or demyelinating) neuropathy, toxic neuropathy (i.e. heavy metal poisoning, drug toxicity, industrial agent exposure), mixed connective tissue disease, severe deforming rheumatoid or osteoarthritis in the limb.
* Conditions that, in the opinion of the study team, may impact the immunomodulatory protocol potentially exposing the recipient to an unacceptable risk under immunosuppressive treatment, including all liver and renal disease.
* Sensitized recipients with high levels (>=50%) of panel-reactive HLA antibodies.
* Conditions that may impact the success of the surgical procedure or increase the risk of postoperative complications including inherited coagulopathies like Hemophilia, Von-Willebrand's disease, Protein C and S deficiency, Thrombocythemias, Thalassemias, Sickle Cell disease, etc.
* Mixed connective tissue diseases and collagen diseases can result in poor wound healing after surgery.
* Conditions that may impact functional outcomes including lipopolysaccharidosis and amyloidosis (may impact nerve regeneration) or rare disorders of bone healing like osteopetrosis.
* Pregnant, breastfeeding or planning to become pregnant within the next 2 years.
* Unable or unwilling to use an acceptable birth control method for 2 years following transplant. The patient cannot have given birth in the past 2 years. We acknowledge that a female recipient of childbearing age must carefully consider the associated risks of the transplant and immunosuppression and personally prioritize these issues and the lead face transplant surgeon (Dr. Cetrulo) will implement this subject in the preoperative education of the patient during consultation.
* Patients will be required to stop smoking for 6 months prior to listing and abstain from postoperative smoking
* If a subject does not receive a transplant after one year of enrollment, clinical consent will be re-obtained from that subject and clinical consent will be re-obtained yearly while the subject is enrolled and waiting for a donor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Incidence of motor function of face | 1 Year
  Function of face as assessed by ability to move face, smile, frown, etc.
Incidence of intact sensation of face | 1 Year
  Sensation of face intact using standard methods (sharp vs dull, presence of numbness)
Incidence of an ascetically satisfactory appearing face | 1 Year
  Evaluated by overall appearance, symmetry
Incidence of a cost benefit to facial transplant | 1 Year
  This will be assessed by standard treatment of facial disfigured patients vs face transplant

SECONDARY OUTCOMES:
Incidence of rejection episodes on triple therapy immunosuppression | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Curt Cetrulo, MD, FACS, FAAP, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No